CLINICAL TRIAL: NCT01503021
Title: A Randomized, Double-Blinded, Placebo-Controlled, Crossover, Multicenter Phase III Safety Study of Soluble Ferric Pyrophosphate (SFP) in Dialysate in Chronic Kidney Disease Patients Receiving Chronic Hemodialysis
Brief Title: Safety Study of Soluble Ferric Pyrophosphate (SFP) in Dialysate in CKD Patients Receiving Chronic Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RMTI-SFP-6
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Results first posted 2015-04-21 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: End Stage Renal Disease; Chronic Kidney Disease
Keywords: Soluble ferric pyrophosphate; Chronic kidney disease; Chronic hemodialysis; Ferric pyrophosphate citrate
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SFP/Placebo (Other): Soluble ferric pyrophosphate (SFP) 2 µmoles (110 µg) iron/L of dialysate in liquid bicarbonate concentrate x 2 weeks, then 1 week washout, then standard liquid bicarbonate concentrate without SFP x 2 weeks
  Interventions: Drug: SFP; Other: Placebo
- Placebo/SFP (Other): Standard liquid bicarbonate concentrate without SFP x 2 weeks, then 1 week washout, then soluble ferric pyrophosphate (SFP) 2 µmoles (110 µg) iron/L of dialysate in liquid bicarbonate concentrate x 2 weeks.
  Interventions: Drug: SFP; Other: Placebo

INTERVENTIONS:
Drug: SFP — Dialysis with SFP administered via the liquid bicarbonate concentrate at a concentration of 2 µmoles (110 µg) iron/L of dialysate
  Other Names: Soluble ferric pyrophosphate
Other: Placebo — Dialysis with standard liquid bicarbonate concentrate without iron
  Other Names: Standard liquid bicarbonate concentrate

SUMMARY:
The purpose of the parent study is to assess the short-term safety and tolerability of soluble ferric pyrophosphate (SFP) in dialysate administered to a large number of representative adult chronic kidney disease patients on hemodialysis (CKD-HD).

The purpose of the extension study is to assess the long-term safety and tolerability of SFP.

DETAILED DESCRIPTION:
Parent Study: randomized, double-blinded, crossover, up to 6 weeks, 700 patients. Patients were randomized to receive SFP 2 µmoles (110 µg) iron/L of dialysate in liquid bicarbonate concentrate or placebo (standard liquid bicarbonate concentrate) x 2 weeks, then a 1 week washout, then crossed over to the alternate treatment x 2 weeks.

Extension Study: open-label, single active arm, uncontrolled study, up to 53 weeks, 300 patients. Following completion of the RMTI-SFP-6 parent study, patients could enter the extension study, where they received SFP 2 µmoles (110 µg) iron/L of dialysate in liquid bicarbonate concentrate for up to 52 weeks.

ELIGIBILITY:
Parent Study, Double Blinded, Crossover:

Key Inclusion Criteria:

1. Adult ≥ 18 years of age.
2. Has chronic kidney disease (CKD) receiving maintenance hemodialysis (HD) (CKD-HD subjects) and regularly undergoing 2 or more dialysis sessions per week.
3. Stable pre-dialysis Hgb ≥ 9.0 to ≤ 12.5 g/dL.
4. Stable pre-dialysis TSAT ≥ 15% to ≤ 45%.
5. Stable pre-dialysis ferritin ≥ 100 to ≤ 1200 µg/L (1200 ng/mL).

Key Exclusion Criteria:

1. Any previous exposure to SFP.
2. Therapy with intravenous, intramuscular or oral iron at any time between the first/screening visit and the randomization visit, or anticipated requirement for iron supplementation during the study period.
3. Non-tunneled vascular catheter for dialysis.
4. Scheduled for kidney transplant within the next 8 weeks.
5. Active infection requiring systemic antimicrobial or antifungal therapy within 2 weeks prior to screening, or during screening period prior to randomization.
6. Hospitalization within 1 month prior to screening (except for vascular access surgery).

Extension Study, Open Label, Single Active Arm:

Key Inclusion Criteria:

1. Participated in Parent Study RMTI-SFP-6 and completed the follow-up/early term visit.
2. Hemoglobin ≤12.0 g/dL at screening.
3. TSAT ≤45% at screening. (Excursion of TSAT by ≤10% outside this range permitted only if all other inclusion/exclusion criteria are met).
4. Serum ferritin ≤1000 µg/L at screening. (Excursion of ferritin by ≤10% outside this range permitted only if all other inclusion/exclusion criteria are met).

Key Exclusion Criteria:

1. Had a serious adverse event attributable (i.e., probably, possibly, or definitely related) to study drug or had an adverse event attributable to study drug that necessitated premature withdrawal from the double-blind, placebo-controlled crossover phase of the parent study RMTI-SFP-6.
2. Non-tunneled vascular catheter for dialysis.
3. Scheduled for kidney transplant within 12 weeks after entry into extension phase.
4. Active infection requiring systemic antimicrobial or antifungal therapy within 2 weeks prior to dosing.
5. Pregnancy or intention to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Pratt, MD, Study Director — Rockwell Medical, Inc
Locations (31):
- United States (28):
  - Mobile, Alabama
  - Northridge, California
  - Arvada, Colorado
  - Westminster, Colorado
  - Lauderhill, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Columbus, Indiana
  - Wichita, Kansas
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Camp Springs, Maryland
  - Gulfport, Mississippi
  - McComb, Mississippi
  - Tupelo, Mississippi
  - City of Saint Peters, Missouri
  - Lincoln, Nebraska
  - Reno, Nevada
  - Rocky Mount, North Carolina
  - Dayton, Ohio
  - Columbia, South Carolina
  - Research Across America, Houston, Texas
  - Houston, Texas
  - Irving, Texas
  - Mission, Texas
  - Temple, Texas
  - Tyler, Texas
- Canada (3):
  - Courtice, Ontario
  - Montreal, Quebec
  - Regina, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SFP/Placebo | Placebo/SFP
Started | 360 | 358
Dosed | 351 | 352
Completed Treatment | 333 | 333 (One patient completed the treatment period but discontinued prior to completing the follow-up visit.)
Completed | 333 | 332
Not Completed | 27 | 26
Not completed — Adverse Event | 7 | 6
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Moved, received transplant, etc. | 5 | 7

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- SFP/Placebo: Soluble ferric pyrophosphate (SFP) 2 µM (110 µg) iron/L of dialysate in liquid bicarbonate concentrate x 2 weeks, then 1 week washout, then standard liquid bicarbonate concentrate without SFP x 2 weeks
- Placebo/SFP: Standard liquid bicarbonate concentrate without SFP x 2 weeks, then 1 week washout, then soluble ferric pyrophosphate (SFP) 2 µM (110 µg) iron/L of dialysate in liquid bicarbonate concentrate x 2 weeks.
- Total: Total of all reporting groups
Arm/Group | SFP/Placebo | Placebo/SFP | Total
Number analyzed (Participants) | 351 | 352 | 703
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (13.18) | 59.5 (13.30) | 59.7 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 141 | 278
  Male | 214 | 211 | 425
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 90 | 106 | 196
  Not Hispanic or Latino | 261 | 246 | 507
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 0 | 5
  Asian | 6 | 8 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 154 | 145 | 299
  White | 185 | 194 | 379
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events
Description: Adverse events for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: percentage of participants
Groups:
- Soluble Ferric Pyrophosphate: Parent Study: Blinded soluble ferric pyrophosphate administered via the liquid bicarbonate concentrate to yield a final dialysate concentration of 2 micromolar (110 micrograms) iron/liter.
- Placebo: Parent Study: Blinded standard liquid bicarbonate concentrate
- Open-label Soluble Ferric Pyrophosphate: Extension Study: Open-label soluble ferric pyrophosphate administered via the liquid bicarbonate concentrate to yield a final dialysate concentration of 2 micromolar (110 micrograms) iron/liter.
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
percentage of participants | 31.6 | 35.1 | 95.1

2. Primary Outcome: Incidence of Treatment-emergent Adverse Events of Intradialytic Hypotension
Description: Adverse events for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. For each adverse event, investigators assessed whether the event met the protocol criteria for intradialytic hypotension. Intradialytic hypotension events were only to have been reported as adverse events if they exceeded the individual subject's baseline pattern of intradialytic hypotension.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: percentage of participants
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
percentage of participants | 4.3 | 4.9 | 12.6

3. Primary Outcome: Incidence of Related Suspected Hypersensitivity Reactions
Description: Adverse events for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. For each adverse event, investigators assessed whether the event met protocol criteria for suspected hypersensitivity reactions.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: percentage of participants
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
percentage of participants | 0 | 0 | 0

4. Secondary Outcome: Incidence of Composite Cardiovascular Events
Description: Adverse events for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. Adverse event terms meeting criteria for composite cardiovascular events were pre-specified in the statistical analysis plan for the study.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: percentage of participants
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
percentage of participants | 1.0 | 0.7 | 13.6

5. Secondary Outcome: Incidence of Hemodialysis Vascular Access Thrombotic Events
Description: Adverse events for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. Adverse event terms meeting criteria for hemodialysis vascular access thrombotic events were pre-specified in the statistical analysis plan for the study.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: percentage of participants
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
percentage of participants | 0.6 | 0.6 | 17.8

6. Secondary Outcome: Incidence of Other Thrombotic Events
Description: Adverse events for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. Adverse event terms meeting criteria for other thrombotic events were pre-specified in the statistical analysis plan for the study.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: percentage of participants
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
percentage of participants | 0 | 0.1 | 1.9

7. Secondary Outcome: Incidence of Systemic/Serious Infections
Description: Adverse events for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. Adverse events of systemic/serious infections were defined in the statistical analysis plan for the study to include infections for which the subject was administered at least 3 doses of an IV antibiotic, and infections for which the subject was hospitalized.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: percentage of participants
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
percentage of participants | 0.4 | 0.9 | 11.3

8. Secondary Outcome: Incidence of Serious Adverse Events
Description: Adverse events for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. For each adverse event, investigators assessed whether the event met seriousness criteria.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: percentage of participants
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
percentage of participants | 4.3 | 5.1 | 46.6

9. Other Pre Specified Outcome: Serum Iron Change From Pre-dialysis to Post-dialysis at Week 2
Description: Serum iron was assessed from samples obtained pre-dialysis and post-dialysis at a single hemodialysis during study week 2. Because of the crossover nature of the study, the week 2 values reflect effects of SFP in the SFP/Placebo arm and effects of Placebo in the Placebo/SFP arm.
Time Frame: Pre-dialysis and post-dialysis during study week 2 of the Parent (Crossover) Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: micromoles per liter
Groups:
- SFP/Placebo: Parent Study: Blinded soluble ferric pyrophosphate (SFP) 2 µmoles (110 µg) iron/L of dialysate, then 1 week washout, then blinded standard liquid bicarbonate concentrate without SFP x 2 weeks
  SFP: Dialysis with SFP administered via the liquid bicarbonate concentrate at a concentration of 2 µmoles (110 µg) iron/L of dialysate
  Placebo: Dialysis with standard liquid bicarbonate concentrate without iron
- Placebo/SFP: Parent Study: Blinded standard liquid bicarbonate concentrate without SFP x 2 weeks, then 1 week washout, then soluble ferric pyrophosphate (SFP) 2 µmoles (110 µg) iron/L of dialysate x 2 weeks.
  SFP: Dialysis with SFP administered via the liquid bicarbonate concentrate at a concentration of 2 µmoles (110 µg) iron/L of dialysate
  Placebo: Dialysis with standard liquid bicarbonate concentrate without iron
Arm/Group | SFP/Placebo | Placebo/SFP
Number analyzed (Participants) | 307 | 311
micromoles per liter
  Pre-dialysis | 13.66 (5.435) | 13.65 (5.299)
  Post-dialysis | 38.60 (10.151) | 14.97 (7.753)
  Change from pre-dialysis to post-dialysis | 24.91 (9.243) | 1.36 (5.447)

10. Other Pre Specified Outcome: Serum Iron Change From Pre-dialysis to Post-dialysis at Week 5
Description: Serum iron was assessed from samples obtained pre-dialysis and post-dialysis at a single hemodialysis during study week 5. Because of the crossover nature of the study, the week 5 values reflect effects of Placebo in the SFP/Placebo arm and effects of SFP in the Placebo/SFP arm.
Time Frame: Pre-dialysis and post-dialysis during study week 5 of the Parent (Crossover) Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | SFP/Placebo | Placebo/SFP
Number analyzed (Participants) | 299 | 303
micromoles per liter
  Pre-dialysis | 12.97 (4.731) | 13.02 (4.856)
  Post-dialysis | 13.98 (7.884) | 37.79 (11.183)
  Change from pre-dialysis to post-dialysis | 1.12 (6.834) | 24.82 (9.827)

11. Other Pre Specified Outcome: Unsaturated Iron-binding Capacity Change From Pre-dialysis to Post-dialysis at Week 2
Description: Unsaturated iron-binding capacity was assessed from samples obtained pre-dialysis and post-dialysis at a single hemodialysis during study week 2. Because of the crossover nature of the study, the week 2 values reflect effects of SFP in the SFP/Placebo arm and effects of Placebo in the Placebo/SFP arm.
Time Frame: Pre-dialysis and post-dialysis during study week 2 of the Parent (Crossover) Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | SFP/Placebo | Placebo/SFP
Number analyzed (Participants) | 351 | 352
micromoles per liter
  Pre-dialysis | 27.95 (6.310) | 28.05 (7.442)
  Post-dialysis | 11.44 (6.899) | 30.49 (8.909)
  Change from pre-dialysis to post-dialysis | -16.47 (7.040) | 2.49 (4.910)

12. Other Pre Specified Outcome: Unsaturated Iron-binding Capacity Change From Pre-dialysis to Post-dialysis at Week 5
Description: Unsaturated iron-binding capacity was assessed from samples obtained pre-dialysis and post-dialysis at a single hemodialysis during study week 5. Because of the crossover nature of the study, the week 5 values reflect effects of Placebo in the SFP/Placebo arm and effects of SFP in the Placebo/SFP arm.
Time Frame: Pre-dialysis and post-dialysis during study week 5 of the Parent (Crossover) Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | SFP/Placebo | Placebo/SFP
Number analyzed (Participants) | 351 | 352
micromoles per liter
  Pre-dialysis | 28.80 (6.745) | 29.05 (7.311)
  Post-dialysis | 30.95 (8.488) | 12.41 (8.463)
  Change from pre-dialysis to post-dialysis | 2.05 (5.333) | -16.68 (7.452)

13. Other Pre Specified Outcome: Transferrin Saturation Change From Pre-dialysis to Post-dialysis at Week 2
Description: Transferrin saturation (based on TIBC derived from transferrin levels) was assessed from samples obtained pre-dialysis and post-dialysis at a single hemodialysis during study week 2. Because of the crossover nature of the study, the week 2 values reflect effects of SFP in the SFP/Placebo arm and effects of Placebo in the Placebo/SFP arm.
Time Frame: Pre-dialysis and post-dialysis during study week 2 of the Parent (Crossover) Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: percent transferrin saturation
Arm/Group | SFP/Placebo | Placebo/SFP
Number analyzed (Participants) | 351 | 352
percent transferrin saturation
  Pre-dialysis | 30.31 (11.357) | 30.46 (11.849)
  Post-dialysis | 80.85 (17.646) | 30.23 (14.397)
  Change from pre-dialysis to post-dialysis | 50.44 (17.442) | -0.25 (10.348)

14. Other Pre Specified Outcome: Transferrin Saturation Change From Pre-dialysis to Post-dialysis at Week 5
Description: Transferrin saturation (based on TIBC derived from transferrin levels) was assessed from samples obtained pre-dialysis and post-dialysis at a single hemodialysis during study week 5. Because of the crossover nature of the study, the week 5 values reflect effects of Placebo in the SFP/Placebo arm and effects of SFP in the Placebo/SFP arm.
Time Frame: Pre-dialysis and post-dialysis during study week 5 of the Parent (Crossover) Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: percent transferrin saturation
Arm/Group | SFP/Placebo | Placebo/SFP
Number analyzed (Participants) | 351 | 352
percent transferrin saturation
  Pre-dialysis | 26.75 (10.302) | 28.88 (10.585)
  Post-dialysis | 28.73 (15.818) | 79.18 (20.008)
  Change from pre-dialysis to post-dialysis | 0.10 (13.792) | 50.42 (18.163)

15. Other Pre Specified Outcome: Ferritin
Description: The baseline and end of treatment predialysis ferritin levels were evaluated for the 52-week extension study to determine whether soluble ferric pyrophosphate increases iron stores.
Time Frame: Baseline, up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 309
micrograms per liter
  Baseline | 653.0 (288.70)
  End of Treatment | 520.3 (341.84)
  Change from Baseline | -132.0 (311.15)

16. Other Pre Specified Outcome: Serum Iron
Description: The baseline and end of treatment predialysis serum iron levels were evaluated for the 52-week extension study to determine the effect of soluble ferric pyrophosphate on serum iron.
Time Frame: Baseline, up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 309
micromoles per liter
  Baseline | 12.650 (4.6488)
  End of Treatment | 11.815 (5.3443)
  Change from Baseline | -0.772 (5.2686)

17. Other Pre Specified Outcome: Transferrin Saturation
Description: The baseline and end of treatment predialysis transferrin saturation were evaluated for the 52-week extension study to confirm clearance of iron derived from soluble ferric pyrophosphate.
Time Frame: Baseline, up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Mean (Standard Deviation); unit: percent transferrin saturation
Arm/Group | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 309
percent transferrin saturation
  Baseline | 30.050 (10.0504)
  End of Treatment | 28.114 (11.5075)
  Change from Baseline | -1.835 (11.7221)

18. Other Pre Specified Outcome: Incidence of Patients Meeting Hy's Law Criteria
Description: The peak alanine aminotransferase and the peak total bilirubin levels were evaluated per patient. Laboratory values for a given intervention (SFP or Placebo) are counted from the date of the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. Patients with alanine aminotransferase more than three times the upper limit of normal and also total bilirubin more than two times the upper limit of normal are counted.
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Population: All participants who received at least one dose of study drug (SFP or placebo, as applicable).
Measure: Number; unit: participants
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Number analyzed (Participants) | 693 | 687 | 309
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 7 weeks for the Parent (Crossover) Study and up to 53 weeks for Extension Study
Description: Adverse events for a given intervention are counted from the first day of dosing of the intervention until 7 days after the last day of dosing of the intervention. Information regarding adverse events was elicited from participants using non-leading questions at each study visit, which generally occurred 3 times per week during the study.
Arm/Group | Soluble Ferric Pyrophosphate | Placebo | Open-label Soluble Ferric Pyrophosphate
Serious Adverse Events (participants affected / at risk) | 30/693 | 35/687 | 144/309
Other Adverse Events (participants affected / at risk) | 123/693 | 131/687 | 253/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Soluble Ferric Pyrophosphate (N=693) | Placebo (N=687) | Open-label Soluble Ferric Pyrophosphate (N=309)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 5
Acute myocardial infarction (Cardiac disorders) | 4 | 1 | 5
Angina pectoris (Cardiac disorders) | 0 | 1 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 4
Cardiac arrest (Cardiac disorders) | 0 | 1 | 4
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 6
Coronary artery disease (Cardiac disorders) | 0 | 2 | 5
Myocardial infarction (Cardiac disorders) | 1 | 3 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2
Gait disturbance (General disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 4
Bronchitis (Infections and infestations) | 0 | 2 | 6
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 5 | 7
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1 | 5
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 3
Syncope (Nervous system disorders) | 2 | 1 | 5
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 3
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 4
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 4
Asthenia (General disorders) | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 2
Medical device complication (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 2
Adverse drug reaction (General disorders) | 0 | 0 | 1
Device pacing issue (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 3
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 6
Cellulitis (Infections and infestations) | 0 | 0 | 5
Gangrene (Infections and infestations) | 0 | 0 | 4
Septic shock (Infections and infestations) | 0 | 0 | 4
Diabetic foot infection (Infections and infestations) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Arteriovenous fistula site infection (Infections and infestations) | 0 | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 2
Abscess limb (Infections and infestations) | 0 | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 0 | 1
Chest wall abscess (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Nasal abscess (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 0 | 1
Areriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 9
Diabetic foot (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 3
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 2
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Steal syndrome (Vascular disorders) | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Retinal artery embolism (Eye disorders) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Soluble Ferric Pyrophosphate (N=693) | Placebo (N=687) | Open-label Soluble Ferric Pyrophosphate (N=309)
Anaemia (Blood and lymphatic system disorders) | 8 | 6 | 20
Diarrhoea (Gastrointestinal disorders) | 9 | 15 | 53
Nausea (Gastrointestinal disorders) | 12 | 12 | 61
Vomiting (Gastrointestinal disorders) | 8 | 8 | 37
Oedema peripheral (General disorders) | 5 | 8 | 36
Upper respiratory tract infection (Infections and infestations) | 4 | 9 | 26
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 11 | 9 | 56
Procedural hypotension (Injury, poisoning and procedural complications) | 32 | 32 | 39
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 15 | 20
Dizziness (Nervous system disorders) | 5 | 7 | 37
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 27
Hypertension (Vascular disorders) | 7 | 5 | 26
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 3 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 32
Fluid overload (Metabolism and nutrition disorders) | 5 | 1 | 18
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 4 | 3 | 49
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4 | 20
Nasopharyngitis (Infections and infestations) | 4 | 1 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 32
Pyrexia (General disorders) | 1 | 1 | 27
Urinary tract infection (Infections and infestations) | 2 | 3 | 21
Vascular graft complication (Injury, poisoning and procedural complications) | 2 | 2 | 27
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 | 3 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less